CLINICAL TRIAL: NCT05815966
Title: The Effect of Emotion Recognition and Empathy Focused Education Program Applied to Earthquake Survivors on Anxiety, Rumination and Post-traumatic Growth Levels of Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gaziantep Islam Science and Technology University (Other)
Collaborators: Duygu Ayar (Unknown); Ayşe Eminoğlu (Unknown)
Responsible Party: Principal Investigator, Ayşe Elkoca, Asist.Prof.Dr. Ayşe Elkoca, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 29-03-2023/ 61
Record Dates: First submitted 2023-03-30; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Anxiety
Keywords: Anxiety; earthquake; fear; rumination; growth after trauma
MeSH Terms: conditions — Anxiety Disorders; Rumination Syndrome

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: emotion recognition and empathy focused training program (Experimental): A suitable hall for children will be determined by the school administration. Education days and hours for the children in the experimental group will be determined by negotiating with the 4th grade teachers. In this study, a 50-minute training program consisting of 2 sessions per week, lasting 5 weeks, will be applied to the experimental group.
  Interventions: Behavioral: The effect of emotion recognition and empathy focused education program
- Control group (No Intervention): Standard care group

INTERVENTIONS:
Behavioral: The effect of emotion recognition and empathy focused education program — Emotion recognition and empathy-oriented education program is a group-based, interactive program that includes techniques such as vision development, brainstorming, painting and drawing, recital, role-playing, gamification and information notes, which requires the active participation of children. Within the program; There are trainings aimed at establishing bilateral relations, gaining in-group commitment, expressing emotions comfortably, feeling that they are not alone, and learning new resources that will make them feel good when they feel bad.
  The aims of education; children,
  Arms: Experimental: emotion recognition and empathy focused training program

SUMMARY:
Earthquakes cause increased mental health problems in the communities they hit. Few attempts have been made to develop effective psychological care strategies for earthquake survivors. Interventions are needed to deal with traumatic stress issues in large populations that survive devastating earthquakes. Fear and anxiety post-traumatic growth and rumination can coexist in individuals after traumatic experiences, and the cognitive pathways leading to them may be different. However, to date, no study has examined the effect of emotion recognition and empathy focused education program on anxiety, rumination and post-traumatic growth levels. This situation constitutes the original value of this project. The aim of this project is to investigate the effect of the emotion recognition and empathy-oriented education program applied to earthquake survivors on children's anxiety, rumination and post-traumatic growth levels. The data of this project, which is planned in accordance with the experimental research principles, will be collected in two primary schools planned to be opened after 13 March 2023. Demographic information form, Event-Related Rumination Inventory, Post-Traumatic Growth Inventory, and Child Anxiety Scale-State and Child Fear Inventory will be used as the project data collection form. The results obtained in this project are planned to be presented as an oral presentation at a national or international congress that will take place in 2023 or 2024 with the theme of child health, nursing or disaster nursing.

The data of the research will be evaluated with the SPSS 20.0 program on the computer. Percentage, mean and t test will be used in the analysis of the data. Chi-square test, Sperman correlation and Wilcoxon test will be used for categorical comparisons. The significance level will be accepted as 0.05 in all statistical processes used within the scope of the research. The significance level will be accepted as 0.05 in all statistical processes used within the scope of the research.

DETAILED DESCRIPTION:
Affecting the health of individuals living in the community mentally, physically and socially; Events that cause death, illness and disability and cause negative consequences are considered disasters. Natural disasters have always had devastating economic, social, medical and public health consequences for people around the world. In the past century, earthquakes that caused loss of life and destruction have occurred in Turkey. Two earthquakes, 7.7 and 7.6, occurred in southeastern Turkey on February 6, 2023, and the earthquakes caused the death of approximately 45 thousand people, the loss of millions of people homeless, the migration to other cities, the loss of their families and relatives, and economic losses. Earthquakes lead to a number of negative psychological consequences such as fear, anxiety and depression, which have the potential to expose survivors to trauma.The earthquake negatively affects not only adults but also children and adolescents. Most affected children have been exposed to a series of extreme stresses such as being trapped, injured, seeing their homes destroyed, and witnessing the injury, suffering or death of others. Compared with adults, children are particularly prone to experience mental problems as a result of traumatic events. Children lack the experience, skills, and resources to independently negotiate issues that may affect their mental health. Children who have experienced a traumatic event such as an earthquake may face situations such as leaving the place where they live as a result of an unexpected situation or losing the people they love and are close to. This situation can lead to the development of feelings such as pessimism and hopelessness about the future in the child. There are many psychological problems such as hopelessness and deterioration in the sense of confidence among the emotional, cognitive and behavioral negative effects of the child after the earthquake. Although studies have reported that survivors of disasters have a high incidence of fear, anxiety, depression and other psychiatric problems, poor recognition of the problems and the inability of detailed clinical assessment of a large affected population should be taken into account. Therefore, it is very important to plan post-earthquake mental health screening and related initiatives. It has been suggested that fear and anxiety are the most common negative outcomes after traumatic events. However, some positive outcomes such as post-traumatic growth (PTD) have also been reported. PSD refers to positive changes as a result of experiencing a traumatic event, such as a sense of strength and wisdom, increased value to friends and family, and a new appreciation for each new day. More importantly, Anxiety, fear, and PTD can coexist in individuals following traumatic experiences, and therefore an important issue is to examine whether Anxiety and PTD share influencing factors. Previous studies have suggested that rumination may play an important role in the development of anxiety and TSD. Repetitive thoughts about the causes and consequences of negative events or mood are called "rumination" and these thoughts can take two forms: temporary and permanent rumination. The former involves a negative focus on trauma-related clues or negative mood, while the latter involves deliberate re-examination and contemplation about the trauma. For most people, ruminations tend to occur soon after the traumatic event, and can persist for a long time. They found that rumination may have different effects on anxiety and PTG, but these studies are cross-sectional and limited in drawing conclusions about a causal relationship. Therefore, the aim of this study is to examine the effects of the emotion recognition and empathy focused education program on the levels of anxiety, PTG and rumination in children living in Gaziantep after the earthquake that occurred on February 6 in the southeast of Turkey and affected 11 cities.

This study will be carried out to determine the effect of the emotion recognition and empathy focused education program applied to earthquake survivors on the anxiety, rumination and post-traumatic growth levels of children.

In accordance with this purpose:

Determining the decrease in the anxiety, fear and rumination levels of the participants (children in earthquake) and the increase in the post-traumatic growth level.

* In measurable expression; A statistically significant decrease was determined in the anxiety, fear and rumination post-test average scores of the participants compared to their pre-test scores,
* Determining a statistically significant increase in the PTG post-test mean scores of the participants (children in the earthquake) compared to their pre-test scores, Place and Time of the Research: The research will be carried out between April 2023 and October 2023 in two Primary Schools in Şahinbey District of Gaziantep Province.

Population and Sample of the Research: The universe of the research consisted of 400 students studying in 4 classes in two Primary Schools located in Şahinbey district of Gaziantep province. In the determination of this age group, it was taken into consideration that the students were at a level that met the skills such as reading comprehension, play, drama, putting oneself in someone else's shoes, and discussion, and were considered the most appropriate age group to be applied by those who developed the scales used.

The sample of the study was calculated over the power analysis made in the G*Power 3.1 program and the variance analysis effect size value in the reference study. 150 In power analysis; The standard deviation was 1, the power value was 80%, and the effect size was 0.6569833, 30 in the experimental group and 30 in the control group, a total of 60 people (df: 58, F: 60). Considering the possibility of students getting sick and leaving, 80 children, 40 of which are in the experimental group and 40 from the control group, will be included in the study by simple random sampling method after stratification of the children whose parents and themselves voluntarily agreed to participate in the study.

The criteria for inclusion of the participants in the sample; children;

* Being able to speak and understand Turkish,
* The children and their parents have voluntarily given their consent to the research,
* Absence of physical or mental disability,
* Having experienced the February 6 earthquake, Exclusion and Exclusion Criteria;
* Existence of physical and mental disability,
* Having a diagnosis of neurological disease,
* Lack of attention,
* Not attending 1 session,
* Failure to fill one of the scales applied in the tests.

ELIGIBILITY:
Inclusion Criteria:

* Being able to speak and understand Turkish,
* The children and their parents have voluntarily given their consent to the research,
* Absence of physical or mental disability,
* Having experienced the February 6 earthquake,

Exclusion Criteria:

* Existence of physical and mental disability,
* Having a diagnosis of neurological disease,
* Lack of attention,
* Not attending 1 session,
* Failure to fill one of the scales applied in the tests.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
the Event Related Rumination Inventory | Change in rumination at 5 weeks
  This scale was developed to measure intrusive and voluntary ruminations after traumatic events and consists of 20 items in total for both types of rumination. In the first part of the scale, there are 10 questions in which participants are asked to indicate how much the event occupied them, even though they try not to think about the traumatic experience, and these questions measure the level of intrusive rumination. The questions in the second part, on the other hand, determine the level of voluntary rumination through the answers given to how much thought of the event, especially and intentionally, after the traumatic experience. The scale is scored as a 4-point Likert scale. In the validity and reliability study of the scale, it is stated that the internal consistency scores are strong and explain 57% of the variance.A minimum of 0 points and a maximum of 60 points are taken from the scale.A high score on the scale indicates that repetitive thoughts about the event increase.
Child Anxiety Scale-State Scale | Change in anxiety at 5 weeks
  It is similar to a thermometer with a light bulb at the bottom and horizontal lines at intervals that go up. This scale, for children aged 4-10, is instructed to "Imagine all anxious or angry feelings are at the bottom here (point to the scale)". If you're a little worried or nervous, the emotions may be a little heightened (put your finger up). If you are very, very anxious or nervous, the emotions may run high (move your finger to the top). The use of the scale is explained as "Put a line showing how anxious or angry you feel". To measure the child's state anxiety, the child is asked to mark what he feels "at the moment". Before the children fill out the ÇAS-D scale, the child's sequencing ability is monitored. A transparent meter is placed above the child's rating with 0.5 point increments marked, then 0.5 point increments are rounded up to the nearest number. The score can vary between 0-10.
Child Fear Scale | Change in fear at 5 weeks
  It is used to measure the child's fear level. The CDS is a scale of 0-4, consisting of showing five drawn facial expressions ranging from neutral (0=no fear) to frightened face (4=severe fear). The fear experienced by the child before, during and after the procedure can be used in the evaluation by parents or researchers. The scale is intended for children aged 5-10 years.
Post Traumatic Growth Scale | Change in post traumatic growth at 5 weeks
  This 21-item scale was developed by Tedeschi and Calhoun (1996) to evaluate the positive development/transformations that can be seen in individuals after traumatic experiences. This scale was translated into Turkish by Dirik (2006) considering the Kılıç (2005) translation. In this study, it was used to evaluate the positive transformations that may occur after trauma and to investigate the factors that contribute to positive results. Using the translation of Dirik (2006) and the 5-factor structure.Posttraumatic growth (PTG) total score (Mean = 2.81, SD = 1.23, Min = 0, Max = 5, Range = 5) was calculated by summing the responses to 21 items and dividing by the number of items. A high mean score indicates greater development after a traumatic experience.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Elkoca, Study Director — Gaziantep Islam Science and Technology University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu J, Xie L, Li B, Li N, Yang Y. Anxiety symptoms among children after the Wenchuan earthquake in China. Nord J Psychiatry. 2012 Oct;66(5):349-54. doi: 10.3109/08039488.2011.650197. Epub 2012 Jan 30. PMID 22283715
- [Background] Dutta A, Pena F, Holcomb JM, Leiva L, Squicciarini AM, Canenguez KM, Bergmann P, Riobueno-Naylor A, Farley AM, Simonsohn A, Garfin DR, Cohen Silver R, Benheim TS, Guzman J, Jellinek MS, Murphy JM. Earthquake exposure, adverse childhood experiences, and psychosocial functioning in Chilean children: A longitudinal study. J Trauma Stress. 2022 Aug;35(4):1177-1188. doi: 10.1002/jts.22826. Epub 2022 Mar 30. PMID 35355336
- [Background] Forresi B, Caputi M, Scaini S, Caffo E, Aggazzotti G, Righi E. Parental Internalizing Psychopathology and PTSD in Offspring after the 2012 Earthquake in Italy. Children (Basel). 2021 Oct 17;8(10):930. doi: 10.3390/children8100930. PMID 34682196